CLINICAL TRIAL: NCT06665737
Title: A Comparison Outcomes of Early and Late Administration G-CSF for Primary Prophylaxis in Non-Hodgkin's Lymphoma Patients Who Receive Chemotherapy, Multicenter Study
Brief Title: Outcomes of Early and Late Administration G-CSF for Primary Prophylaxis in Non-Hodgkin's Lymphoma Patients
Acronym: G-CSF in NHL
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Mahidol University (Other); Internal Medicine Unit, Pranangklao Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205/2567; Rajavithi Hospital (Other Grant/Funding Number: Rajavithi Hospital)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-10

CONDITIONS: Non-Hodgkin's Lymphoma (NHL); Granulocyte Colony Stimulating Factor; Febrile Neutropenia (FN); Myelosuppression Adult
Keywords: Non-Hodgkin's lymphoma; Febrile neutropenia; Granulocyte Colony Stimulating Factor; Myelosuppression
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Febrile Neutropenia

STUDY DESIGN:
Intervention Model Description: Group A: Early receiving G-CSF Group B: Late receiving G-CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early receiving G-CSF group (Active Comparator): Early receiving G-CSF group Patients in early receiving G-CSF group accept within 72 hours post chemotherapy
  Interventions: Drug: Early receiving G-CSF group
- Late receiving G-CSF group (Placebo Comparator): Last receiving G-CSF group Patients in early receiving G-CSF group accept after 72 hours post chemotherapy
  Interventions: Drug: Late receiving G-CSF group

INTERVENTIONS:
Drug: Early receiving G-CSF group — Early receiving G-CSF group will be given within 72 hours post chemotherapy
  Arms: Early receiving G-CSF group
Drug: Late receiving G-CSF group — Late receiving G-CSF group will be given after 72 hours post chemotherapy
  Arms: Late receiving G-CSF group

SUMMARY:
The goal of this clinical trial is to

Primary Objectives:

1. To compare the incidence of febrile neutropenia in patients with non-Hodgkin's lymphoma who received early or late granulocyte colony-stimulating factor (G-CSF) during standard chemotherapy in a multicenter study
2. To determine the incidence of leukopenia and neutropenia in patients with non-Hodgkin's lymphoma who received early or late G-CSF during standard chemotherapy in a multicenter study

Secondary Objectives:

1. To determine changes in white blood cell, hemoglobin, and platelet levels in patients with non-Hodgkin's lymphoma who received early or late G-CSF during standard chemotherapy.
2. To determine the quality of life of patients with non-Hodgkin's lymphoma who undergoing standard chemotherapy and with neutropenia Researchers will compare the outcome between patients received either early G-CSF (within 72 hours) or late G-CSF (after 72 hours).

All patients will be followed up to monitor for febrile neutropenia events, other hematological parameters and quality of life.

DETAILED DESCRIPTION:
This study aims to analyze the impact of the timing of granulocyte colony-stimulating factor (G-CSF) administration on the prevention of febrile neutropenia (FN) in non-Hodgkin's lymphoma patients undergoing standard chemotherapy. G-CSF is a growth factor that stimulates the production of white blood cell in order to fighting infection. When non-Hodgkin's lymphoma patients receive chemotherapy for eradicating cancer cells. They also have collateral damage those white blood cells and other hematopoietic cell lines.

All patients received standard chemotherapy regimens once every four weeks. The study will compare the efficacy of early G-CSF administration, or late administration, after each course of chemotherapy.

The primary endpoint is the incidence of FN in each chemotherapy course. At the end of each chemotherapy course, patients received either early G-CSF (within 72 hours) or late G-CSF (after 72 hours). All patients will be followed up to monitor for FN events.

Secondary endpoints include the incidence of myelosuppression and quality of life, assessed during outpatient and emergency department visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or old
* Confirmed lymphoma undergoing standard chemotherapy
* Signed an approval informed consent
* Has a good understanding of Thai
* Available for follow-up after chemotherapy

Exclusion Criteria:

* Pregnancy or lactation
* Serious concomitant diseases and discontinuous treatment such as cardiovascular, liver, or kidney diseases
* Contraindication to chemotherapy or G-CSF administration
* Antibiotic use within 1 week prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia | One year
  Incidence of febrile neutropenia in each course
Incidence of leukopenia and neutropenia | One year
  Incidence of leukopenia and neutropenia in each course

SECONDARY OUTCOMES:
Incidence of grade 3 or 4 of myelosuppression | One year
  Incidence of 3 or 4 myelosuppression in each course
Time of visits to outpatient (OPD) and emergency clinics (ER) | One year
  Incidence of visit to OPD or ER in each course
Quality of life (QoL) after chemotherapy | One year
  Quality of life score daily in each course

CONTACTS AND LOCATIONS:
Locations (3):
- Thailand (3):
  - Department of Clinical Tropical Medicine, Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok
  - Rajavithi Hospital, Bangkok, Bangkok
  - Internal Medicine Unit, Pranongklao Hospital, Nontaburi, Nontaburi

IPD SHARING:
Plan to Share IPD: Undecided